CLINICAL TRIAL: NCT01447771
Title: Decision Support for Women With Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds to continue and volunteer recruitment member left position
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: NA00046799; J1158 (Other: The Sidney Kimmel Comprehensive Cancer Center)
Record Dates: First submitted 2011-09-21; First posted 2011-10-06 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Breast Neoplasms
Keywords: Decision making; Decisional aide
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental): Decision control preference intervention
  Interventions: Behavioral: Decision control preference scale

INTERVENTIONS:
Behavioral: Decision control preference scale — At time 1, participants in the intervention group will be asked to complete the Decision Control Preference Scale.The range of decision control is measured by the Decision Control Preference (DCP) Scale. The scale is used to measure the preferred or actual role in decision making using five response statements: two represent an active or patient-controlled role, one a shared or collaborative role, and two represent a passive or provider-controlled role. The preferred level of decision making control will be known by the participant in the intervention group and the information given to the oncologist prior to the consultation regarding adjuvant therapy
  Other Names: DCP scale

SUMMARY:
Breast cancer is a common malignancy among women in the United States. There are a variety of treatment decisions that need to be made. This study has been developed after a review of the literature demonstrated that women with breast cancer are making decisions regarding complex therapy issues in a way that is not congruent with their decision-making control preference.

Some patients want to be empowered with information so that they can actively participate in the decision making about their care; others want to rely on the recommendations made by the oncologist. This is important because patients who were not satisfied with their adjuvant treatment decision noted a negative effect on quality of life and self image. These patients had more difficulties with treatment side effects; including aches, hot flashes, pain, and mood alteration. In additions the Institute of Medicine recommended that patient centeredness be a key aim of health care organizations and that all patients be given the opportunity to exercise the degree of control they choose over health care decisions that affect them.

It is hypothesized that women making decisions regarding adjuvant therapy who are supported to make decisions based on their preferred level of control will have positive psychological outcomes.

DETAILED DESCRIPTION:
This evidence based study has been developed after a review of the literature demonstrated that 14 - 58% of women with breast cancer are making decisions regarding complex therapy issues in a way that is not congruent with their decision-making control preference. Because of the prevalence of decision-making control preference incongruence and strong evidence that providing support for a woman's decision making control preference is related to quality of life measures, this study will test the implementation of a nursing intervention to support the decision making of women with breast cancer. Using sample randomization with assignment to one of two groups, this study will explore whether using Degner's Control Preference (DCP) Scale supports decision making control preferences in women who are making decisions about breast cancer treatment. Results of the study will guide implementation of sustainable evidence-based behavioral practices that can have significant effects on quality of care outcomes.

This study will assess satisfaction with decision involvement, depression, and decision making distress in women with early stage breast cancer after a decision support intervention to support a woman's preferred decision control preference. It is hypothesized that a decision support intervention that consists of providing information from the Degner Control Preference (DCP) Scale to the provider and patient will have a positive effect on psychological outcomes (decision satisfaction, decision making distress, and depression) in women making decisions about breast cancer treatment. Testing the effect of the decision support intervention on decision satisfaction, decision making distress and depression will be measured using t-Tests.

Patients with early stage breast cancer who are scheduled to have a medical oncology consultation, to decide an adjuvant therapy regimen, will be asked to participate.

128 patients will be randomly assigned to a group in which the patient and their oncologist would know the patient's preferred level of decision making control (intervention group) or a group that would receive information about a balanced diet (attention control group). Two nurses on the research team will consent participants, participate in the intervention, and collect data through interviews. Post intervention interviews will occur within 24 hours of the intervention and 4 weeks later.

ELIGIBILITY:
Inclusion Criteria:

1. Women with early stage (Stage I and Stage II) breast cancer that are considering adjuvant therapy and are being evaluated at the Johns Hopkins Avon Foundation Breast Center.
2. Age 18 years and older.
3. Able to read and speak English.

Exclusion Criteria:

1. Severe visual impairments that would make it difficult to read study instruments or inability to read.
2. Lack of capacity to provide informed consent to participate in the study.
3. Patients being seen for a second opinion.
4. Patients with a history of previous neoadjuvant chemotherapy.
5. Women who are pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Satisfaction with Decision at 24 hours | 24 hours after consultation
  Satisfaction with Decision (SWD) scale: A 6 item tool with a 5-point Likert scale ranging from 1, "strongly disagree" to 5, "strongly agree", will be used to evaluate the patient's satisfaction with decision involvement by phone within 24 hours following the consultation and repeated 4 weeks later. This instrument is based on the Satisfaction with Decision Instrument of Holmes-Rovner. The SWD scale performed reliability, Cronbach's alpha = 0.86
Satisfaction with Decision at 4 weeks | 4 weeks after consultation
  Satisfaction with Decision (SWD) scale: A 6 item tool with a 5-point Likert scale ranging from 1, "strongly disagree" to 5, "strongly agree", will be used to evaluate the patient's satisfaction with decision involvement by phone within 24 hours following the consultation and repeated 4 weeks later. This instrument is based on the Satisfaction with Decision Instrument of Holmes-Rovner. The SWD scale performed reliability, Cronbach's alpha = 0.86

SECONDARY OUTCOMES:
Baseline Depression Score | Baseline before consultation
  This scale will be used to measure depressive symptoms. The CSES-D 10 is a 10-item brief version of a self-report questionnaire developed by the Center for Epidemiologic Studies at the National Institute of Mental Health for use in studies of depression in community samples. The CSES-D 10 version has been used across multiple populations. It has been shown to have test-retest reliability of 0.80 in patients with GI cancer.
Baseline Impact of Event Score | Baseline, before consultation
  A 15-item Likert scale ranging from total scores of 0 to 75 with levels of: 9-25 indicative of moderate adaptation difficulties and > 26 is considered indicative of clinical adaptation difficulties. Intrusion (the extent to which individuals are overwhelmed by thoughts and feelings of breast cancer, 7 items) and avoidance (the tendency to avoid thoughts and feelings about breast cancer, 8 items) are subscales. In this study, it will be used to measure patient distress in participating in health care decision making. The Cronbach's alpha for patients with GI cancer was 0.86.
Depression Score at 4 weeks | 4 weeks after consultation
  This scale will be used to measure depressive symptoms. The CSES-D 10 is a 10-item brief version of a self-report questionnaire developed by the Center for Epidemiologic Studies at the National Institute of Mental Health for use in studies of depression in community samples. The CSES-D 10 version has been used across multiple populations. It has been shown to have test-retest reliability of 0.80 in patients with GI cancer.
Impact of Event score at 24 hours | 24 hours after consultation
  A 15-item Likert scale ranging from total scores of 0 to 75 with levels of: 9-25 indicative of moderate adaptation difficulties and > 26 is considered indicative of clinical adaptation difficulties. Intrusion (the extent to which individuals are overwhelmed by thoughts and feelings of breast cancer, 7 items) and avoidance (the tendency to avoid thoughts and feelings about breast cancer, 8 items) are subscales. In this study, it will be used to measure patient distress in participating in health care decision making. The Cronbach's alpha for patients with GI cancer was 0.86.
Impact of Event Score at 4 weeks | 4 weeks after consultation
  A 15-item Likert scale ranging from total scores of 0 to 75 with levels of: 9-25 indicative of moderate adaptation difficulties and > 26 is considered indicative of clinical adaptation difficulties. Intrusion (the extent to which individuals are overwhelmed by thoughts and feelings of breast cancer, 7 items) and avoidance (the tendency to avoid thoughts and feelings about breast cancer, 8 items) are subscales. In this study, it will be used to measure patient distress in participating in health care decision making. The Cronbach's alpha for patients with GI cancer was 0.86.
Congruence between preferred and actual decision making control at 24 hours | 24 hours after consultation
  This is a yes/no answer to determine congruence between actual and preferred level of decision making control. Descriptive analysis of the results will be preformed
Congruence between preferred and actual decision making control at 4 weeks | 4 weeks after consultation
  This is a yes/no answer to determine congruence between actual and preferred level of decision making control. Descriptive analysis of the results will be preformed
Baseline Impact of Event Score | Before consultation
  A 15-item Likert scale ranging from total scores of 0 to 75 with levels of: 9-25 indicative of moderate adaptation difficulties and > 26 is considered indicative of clinical adaptation difficulties. Intrusion (the extent to which individuals are overwhelmed by thoughts and feelings of breast cancer, 7 items) and avoidance (the tendency to avoid thoughts and feelings about breast cancer, 8 items) are subscales. In this study, it will be used to measure patient distress in participating in health care decision making. The Cronbach's alpha for patients with GI cancer was 0.86.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Olsen, PhD, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Degner LF, Kristjanson LJ, Bowman D, Sloan JA, Carriere KC, O'Neil J, Bilodeau B, Watson P, Mueller B. Information needs and decisional preferences in women with breast cancer. JAMA. 1997 May 14;277(18):1485-92. PMID 9145723
- [Background] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581
- [Background] Holmes-Rovner M, Kroll J, Schmitt N, Rovner DR, Breer ML, Rothert ML, Padonu G, Talarczyk G. Patient satisfaction with health care decisions: the satisfaction with decision scale. Med Decis Making. 1996 Jan-Mar;16(1):58-64. doi: 10.1177/0272989X9601600114. PMID 8717600
- [Background] Lo SS, Mumby PB, Norton J, Rychlik K, Smerage J, Kash J, Chew HK, Gaynor ER, Hayes DF, Epstein A, Albain KS. Prospective multicenter study of the impact of the 21-gene recurrence score assay on medical oncologist and patient adjuvant breast cancer treatment selection. J Clin Oncol. 2010 Apr 1;28(10):1671-6. doi: 10.1200/JCO.2008.20.2119. Epub 2010 Jan 11. PMID 20065191
- [Background] Hack TF, Degner LF, Watson P, Sinha L. Do patients benefit from participating in medical decision making? Longitudinal follow-up of women with breast cancer. Psychooncology. 2006 Jan;15(1):9-19. doi: 10.1002/pon.907. PMID 15669023
- [Background] Shaha M, Cox CL, Talman K, Kelly D. Uncertainty in breast, prostate, and colorectal cancer: implications for supportive care. J Nurs Scholarsh. 2008;40(1):60-7. doi: 10.1111/j.1547-5069.2007.00207.x. PMID 18302593